CLINICAL TRIAL: NCT07293078
Title: Prospective Evaluation of a Point-of-Care Artificial Intelligence Model in Critical Care Outcomes
Brief Title: Point-of-Care AI Assistance and Critical Care Outcomes: A Randomized Trial
Acronym: POC-AI-ICU
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MetroWest Artificial Intelligence Research Workgroup (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POC-AI-ICU-001; IRB#2025-067 (Other: MetroWest Medical Center and St. Vincent Hospital)
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Sepsis; Acute Respiratory Failure (ARF); Multi-organ Failure; Acute Kidney Injury; Delirium Confusional State; Shock
Keywords: Critical Care; Intensive Care Unit; Large Language Model; Artificial Intelligence; Diagnostic Accuracy; Clinical Decision Support; Critical Care Outcomes; Sepsis; Shock; Acute Respiratory Failure; Multiorgan Failure
MeSH Terms: conditions — Critical Illness; Sepsis; Multiple Organ Failure; Acute Kidney Injury; Confusion; Shock

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Patients receive usual ICU care per local practice. De-identified admission data may be processed and submitted to the LLM for research purposes, but AI output is not shared with treating clinicians and does not influence real-time management.
- AI-Assisted Care (Other): Patients receive standard ICU care plus point-of-care LLM-based decision support at admission. De-identified admission data are formatted and submitted to an LLM (ChatGPT-5). The model returns a primary diagnosis, ranked differential diagnosis list, suggested additional information, and prioritized therapeutic recommendations. This output is provided to the admitting team for consideration in ongoing management.
  Interventions: Other: Point-of-care large language model decision support (ChatGPT-5)

INTERVENTIONS:
Other: Point-of-care large language model decision support (ChatGPT-5) — Use of a large language model (ChatGPT-5) to analyze de-identified ICU admission data (history, physical examination, laboratory results, imaging reports, and other documentation) at the time of admission. The model generates diagnostic and therapeutic recommendations that are shared with clinicians in the AI-assisted arm only.
  Arms: AI-Assisted Care

SUMMARY:
This is a prospective, unmasked, randomized, multicenter clinical trial evaluating the impact of point-of-care large language model (LLM)-based decision support on diagnostic accuracy and clinical outcomes in adult medical intensive care unit (MICU) patients.

Consecutive adult ICU admissions at participating community hospitals (initially MetroWest Medical Center and St. Vincent Hospital) will be screened for eligibility. Eligible patients will be randomized 1:1 to standard care or an AI-assisted group. In both arms, initial evaluation and management will follow usual practice. For patients randomized to AI assistance, de-identified admission data (history and physical, labs, imaging reports, and other relevant documentation) will be formatted and submitted to a state-of-the-art LLM (ChatGPT-5) at the time of admission. The AI-generated differential diagnosis and therapeutic recommendations will be provided to the admitting team for consideration. For the standard care arm, LLM output will be generated but not shared with clinicians.

After discharge, a masked chart review will determine the "ground truth" primary diagnosis and extract outcomes including: Primary Outcome - a composite of medical errors (from time of ICU admission through day 7 of ICU stay, or ICU discharge, whichever comes first); Secondary Outcomes - 90-day mortality, ICU and hospital length of stay, and ventilator-free days.

DETAILED DESCRIPTION:
The rapid development of large language models (LLMs) such as ChatGPT has created new opportunities and risks for their use in medicine. Although early studies suggest high diagnostic accuracy in complex clinical scenarios and ICU admissions, the impact of LLMs on real-world clinical outcomes and the optimal mode of physician-AI interaction remain uncertain. Published work from our group showed that ChatGPT-4 achieved diagnostic accuracy comparable to board-certified intensivists for ICU admissions in a retrospective study. However, prospective, randomized data on clinical outcomes are lacking.

This trial will evaluate a pragmatic paradigm for integrating LLMs at the time of ICU admission (point-of-care AI). All eligible adult MICU admissions at participating sites will be prospectively randomized to: (1) standard care, or (2) AI-assisted care in which an LLM receives standardized, de-identified admission data and returns a proposed primary diagnosis, ranked differential diagnosis (up to five conditions), suggested additional information, and prioritized therapeutic interventions. Admitting clinicians in the AI-assisted arm will be asked to review and optionally incorporate the AI recommendations and will complete a brief questionnaire regarding perceived utility and any changes in diagnosis or management.

A masked clinical adjudication panel will perform longitudinal chart review to define the "ground truth" primary diagnosis and assess error rates and outcomes. The primary endpoint is a composite of medical errors. The specific time frame will be from the time of ICU admission through day 7 of ICU stay, or ICU discharge, whichever comes first. Secondary endpoints will include 90-day mortality, ICU and hospital length of stay, and ventilator-free days. Other exploratory secondary endpoints will be considered. The trial is designed to enroll approximately 1000 patients across multiple MICUs, with interim analysis at 12 months to assess feasibility, integrity, and futility. The study is minimal risk, uses de-identified data for AI queries, and does not alter standard diagnostic testing or therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years) admitted to the medical intensive care unit (MICU) at participating hospitals.
2. Direct admissions from the emergency department or transfers from medical wards to the MICU.
3. Critically ill patients meeting local ICU admission criteria.

Exclusion Criteria:

1. Transfers to the MICU from outside hospitals, operating room, or post-anesthesia care unit.
2. Age < 18 years.
3. Incomplete or missing essential clinical information at admission (e.g., key labs or documentation not yet available).
4. Primary surgical or cardiac (e.g., STEMI) patients.
5. Pregnant or postpartum women.
6. Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of Medical Errors | From the time of ICU admission through day 7 of ICU stay or ICU discharge, whichever comes first.
  Proportion of patients with at least one clinically important diagnostic or therapeutic error identified by masked chart review (e.g., missed or delayed critical diagnosis, major guideline-discordant therapy with potential for harm).

SECONDARY OUTCOMES:
90-day All-Cause Mortality | 90 days from ICU admission.
  All-cause mortality within 90 days of index ICU admission, as determined by chart review and available follow-up records.
ICU Length of Stay | From ICU admission to ICU discharge (up to 90 days).
  Total number of days spent in the ICU during the index hospitalization.
Ventilator-Free Days | Up to 28 days after ICU admission.
  Number of days alive and free from invasive mechanical ventilation during the first 28 days after ICU admission.
Hospital Length of Stay | From hospital admission to hospital discharge (up to 90 days).
  Total number of days from hospital admission to hospital discharge during the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Silverman, M.D., Principal Investigator — MetroWest Medical Center and St. Vincent Hospital
Locations (1):
- Framingham Union Hospital/MetroWest Medical Center, Framingham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be retained for reanalysis by the study team. There is no current plan for routine public sharing of individual participant-level data, but de-identified datasets may be shared with qualified investigators upon reasonable request and appropriate data use agreements.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Singh J, Bohra R, Mukhtiar V, Fernandes W, Bhanushali C, Chinnamuthu R, Kanamgode SS, Ellis J, Silverman E. Diagnostic Accuracy of a Large Language Model (ChatGPT-4) for Patients Admitted to a Community Hospital Medical Intensive Care Unit: A Retrospective Case Study. J Intensive Care Med. 2025 Aug 17:8850666251368270. doi: 10.1177/08850666251368270. Online ahead of print. PMID 40820407